CLINICAL TRIAL: NCT04164446
Title: Supplementation of Oil Palm Phenolics to Improve Lipid Profile in Healthy Participants (Phase I Clinical Trial Study)
Brief Title: Supplementation of Oil Palm Phenolics to Healthy Participants
Acronym: SPIRAL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Principal Investigator, Isa Naina Mohamed, Associate Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SPIRAL
Record Dates: First submitted 2019-11-10; First posted 2019-11-15 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Diseases; Hyperlipidemias; Hypercholesterolemia
Keywords: oil palm phenolics; lipid profile; LDL cholesterol; HDL cholesterol
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Two capsules containing starch and glucose, once per day, 60 days duration
  Interventions: Drug: Placebos
- Oil Palm Phenolics 250 mg (Active Comparator): One capsule 250 mg active compound (OPP) and one capsule containing starch and glucose, once per day, 60 days duration
  Interventions: Dietary Supplement: Oil Palm Phenolics
- Oil Palm Phenolics 1000 mg (Active Comparator): One capsule containing 1000 mg active compound (OPP) and one capsule starch and glucose, once per day, 60 days duration
  Interventions: Dietary Supplement: Oil Palm Phenolics
- Oil Palm Phenolics 2000 mg (Active Comparator): Two capsules, 1000 mg active compound (OPP) each, once per day, 60 days duration
  Interventions: Dietary Supplement: Oil Palm Phenolics

INTERVENTIONS:
Drug: Placebos — The placebo that will be used contains starch and glucose.
  Other Names: Placebo
  Arms: Placebo
Dietary Supplement: Oil Palm Phenolics — One capsule contains 250 mg OPP or 1 g OPP
  Arms: Oil Palm Phenolics 1000 mg; Oil Palm Phenolics 2000 mg; Oil Palm Phenolics 250 mg

SUMMARY:
Our previous study has found that oil palm phenolics (OPP) supplementation at 9 grams per day is safe for consumption. An interesting observation was reported where the consumption of OPP showed significantly lower total and LDL cholesterol compared to the control group. There is no clinical evidence as yet on the optimum dosage of OPP supplementation in improving fasting lipid profile. We hypothesize that in a clinical study, OPP supplemented participants will elicit a reduction in total and LDL cholesterol while maintaining safety and tolerability.

DETAILED DESCRIPTION:
During the palm oil milling process, a large amount of vegetation liquor is discarded into the aqueous waste stream. A novel process to recover phenolic compounds from the aqueous waste stream were developed and resulting in producing a filtrate known as oil palm phenolics (OPP), which contains a high amount of phenolic. It has been postulated that phenolic acids components found in the OPP have promising health benefits such as antioxidant, anti-inflammatory, neuroprotective and anti-tumour effects.

Hyperlipidemia, one of the risk factors for cardiovascular diseases (CVD), is defined as elevations of fasting total cholesterol or triglyceride concentration or both. Through our current research, OPP supplementation to hamster animal model has shown positive effects in the reduction of total cholesterol and triglycerides as well as improvement of high-density lipoprotein cholesterol (HDL-C). In a previous study using the rabbit animal model, OPP has shown a protective effect against atherosclerosis, a condition whereby fat and cholesterol plaques are deposited inside the arteries. Based on the current evidence from the preliminary studies on OPP, we hypothesize that supplementation of OPP may prevent or delay the development of CVD.

However, to understand the anti-hyperlipidemic effects of OPP in humans, we need to establish our knowledge of the physiological effects of this compound to normal human subjects. Under physiological condition, OPP may improve the antioxidant and anti-inflammatory status. These improvements may have a positive influence on plasma lipid profile since many scientific evidences demonstrate that antioxidant and anti-inflammatory effects may contribute protection against the incidence of CVD. Therefore, we proposed a clinical trial to evaluate the antioxidant and anti-inflammatory effects of OPP in eliciting the possible mechanism for lipid reduction.

This study will be started with the recruitment of 100 healthy volunteers where they will be supplemented with placebo/OPP capsules at different doses for 60 days. Participants will be required to take the placebo/OPP capsules in front of the study staff to ensure compliance. Blood samples will be withdrawn at baseline, day 30 and day 60, and will be analyzed for lipid profile, antioxidant and anti-inflammatory status. Data from this study would hopefully assist us in understanding the therapeutic roles of OPP on humans under normal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal Total Cholesterol level of less than 5.2 mmol/dL
* Normal LDL Cholesterol level of less than 3.36 mmol/dL
* Normal Triglyceride level of less than 1.69 mmol/dL

Exclusion Criteria:

* Smoking
* Habitual alcohol consumption
* Consuming antioxidant supplement
* Pregnant/ breastfeeding
* Medical history of cardiovascular disease, diabetes, dyslipidemia
* Current use of antihypertensive or lipid-lowering medication

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Fasting Plasma LDL Cholesterol level following one and two months supplementation | Baseline, day 30, day 60
  This will be assessed from the plasma analysis on the fasting blood samples of each participant
Incidence of Adverse Events following one-month supplementation (Safety and Tolerability) | Day 30 after supplementation
  This will be assessed via history, physical examination, kidney function test, liver function test and hematology profile from the plasma analysis on the fasting blood samples of each participant.
Incidence of Adverse Events following two-months supplementation (Safety and Tolerability) | Day 60 after supplementation
  This will be assessed via history, physical examination, kidney function test, liver function test and hematology profile from the plasma analysis on the fasting blood samples of each participant.

SECONDARY OUTCOMES:
Changes from Baseline Fasting Lipid Profile (total and HDL cholesterol, triacylglycerides) following one and two months supplementation | Baseline, day 30 and day 60 after supplementation
  This will be assessed from the plasma analysis on the fasting blood samples of each participant.
Changes from Baseline Fasting LDL and HDL Cholesterol Subfractions following one and two months supplementation. | Baseline, day 30 and day 60 after supplementation
  This will be assessed from the plasma analysis on the fasting blood samples of each participant.
Changes from Baseline Concentrations of Plasma Inflammatory Markers using multiplex assays following one and two months supplementation | Baseline,day 30 and day 60 after supplementation
  Inflammatory markers such as Interleukin-6, Interleukin-1beta, Tumour Necrosis Factor-alpha, Interleukin-10 and interferon-Gamma will be assessed from the plasma analysis on the fasting blood samples of each participant.
Changes from Baseline Concentrations of Plasma Antioxidant Levels using ELISA method following one and two months supplementation | Baseline,day 30 and day 60 after supplementation
  Antioxidant levels such as Malonaldehyde and Superoxide dismutase will be assessed from the plasma analysis on the fasting blood samples of each participant.
Changes from Baseline Body Weight Measurement following one and two months supplementation | Baseline,day 30 and day 60 after supplementation
  This will be assessed by measuring the weight of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Isa Naina Mohamed, MD, PhD, Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Cheras, WP Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fairus S, Leow SS, Mohamed IN, Tan YA, Sundram K, Sambanthamurthi R. A phase I single-blind clinical trial to evaluate the safety of oil palm phenolics (OPP) supplementation in healthy volunteers. Sci Rep. 2018 May 29;8(1):8217. doi: 10.1038/s41598-018-26384-7. PMID 29844318
- [Derived] Muhammad Ismail Tadj NB, Ibrahim N', Haji Mohd Saad Q, Tg Abu Bakar Sidik TMI, Leow SS, Fairus S, Naina Mohamed I. A Phase I, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety and Tolerance of Oil Palm Phenolics (OPP) in Healthy Volunteers. Front Pharmacol. 2022 Jun 20;13:893171. doi: 10.3389/fphar.2022.893171. eCollection 2022. PMID 35795564